CLINICAL TRIAL: NCT06539039
Title: The Effect of Non Surgical Periodontal Therapy on the Ratio of TNF-α to IL-10 in Periodontitis Patients With Diabetics Mellites
Brief Title: Periodontal Therapy Effect on the Ratio of TNF-α to IL-10 in Periodontis With/Out DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fDASU-RecIM210223
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Periodontitis Generalized

STUDY DESIGN:
Intervention Model Description: 36 patients with generalized periodontitis, recruited from Ain-Shams University's outpatient clinic. Patients were divided into three groups: poorly controlled diabetes (HbA1c ≥ 7%), controlled diabetes (HbA1c < 7%), and non-diabetic periodontitis. Full-mouth NSPT was performed, and clinical parameters (Plaque Index, Bleeding Index, Pocket Depth, Clinical Attachment Level) were assessed at baseline and eight weeks post-treatment. Venous blood samples were collected to measure TNF-α and IL-10 levels using ELISA kits.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- periodontitis with controlled diabetes (Experimental): patients with generalized periodontitis and controlled diabetes mellitus with glycated haemoglobin (HbA1c) less than 7%.
  Interventions: Procedure: non surgical periodontal therapy
- periodontitis with poorly controlled diabetes (Experimental): patients with generalized periodontitis, and poorly controlled diabetes mellitus with HbA1c more than or equal 7%.
  Interventions: Procedure: non surgical periodontal therapy
- periodontitis (Experimental): patients with generalized periodontitis
  Interventions: Procedure: non surgical periodontal therapy

INTERVENTIONS:
Procedure: non surgical periodontal therapy — participants received full mouth one stage debridement using hand instruments and use of universal curette for sub gingival debridement and ultrasonic scalers through use of supragingival and subgingival ultrasonic tips

SUMMARY:
Periodontitis is a chronic inflammatory disease affecting the periodontium, characterized by irreversible damage to the gingiva, periodontal ligament, and alveolar bone. It is prevalent among adults, significantly impacting oral health and quality of life. This study investigates the effect of non-surgical periodontal therapy (NSPT) on the levels of Tumor Necrosis Factor-alpha (TNF-α) and Interleukin-10 (IL-10) in periodontitis patients with and without diabetes mellitus type II.

DETAILED DESCRIPTION:
A single-blinded, randomized clinical trial was conducted on 36 patients with generalized periodontitis, recruited from Ain-Shams University's outpatient clinic. Patients were divided into three groups: poorly controlled diabetes with periodontitis (HbA1c ≥ 7%), controlled diabetes with periodontitis (HbA1c < 7%), and non-diabetic periodontitis. Full-mouth NSPT was performed, and clinical parameters (Plaque Index, Bleeding Index, Pocket Depth, Clinical Attachment Level) were assessed at baseline and eight weeks post-treatment. Venous blood samples were collected to measure TNF-α and IL-10 levels using ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* Both genders. Age (20-50 ) years old. Participants willing to commit for the entire period of the trial and agreed to sign the written consent after full explanation of the study.

Generalized Periodontitis patients . Having at least 20 tooth excluding wisdoms. Systemically free according to the modified Burkett's health history questionnaire except for diabetes mellitus (Burket, Greenberg and Glick 2003).

Exclusion Criteria:

* Smokers.
* Intake of immunosuppressive drugs, antibiotics or anti-inflammatory drugs throughout the last three months prior to the study .
* status of pregnancy or lactation.
* allergy to local anesthetic.
* Prisoners .
* The vulnerable group ; mentally and physically disabled patients .

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
detect difference in the ratio of tumor necrosis factor-α interleukin-10 in periodontitis patients with and without diabetes | 8 weeks
  To detect difference in the ratio of the proinflammatory cytokine tumor necrosis factor-α to the anti-inflammatory cytokine interleukin-10 between periodontitis patients with and without type 2 diabetes mellitus before and after non surgical periodontal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: mahetab mohamed, lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Dentistry, Cairo, Organization of African Unity St, El-Qobba Bridge, Egypt

IPD SHARING:
Plan to Share IPD: No